CLINICAL TRIAL: NCT06944951
Title: Post-Marketing Clinical Follow-Up Trial to Evaluate the Performance and Safety of the Medical Device PROCTOeze® PLUS in the Relief of Haemorrhoidal Disease and Anal Irritation Symptoms
Brief Title: Post-Marketing Clinical Follow-Up Trial to Evaluate the Performance and Safety of PROCTOeze® PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biokosmes Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OpBio/0123/MD
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Haemorrhoidal Disease
Keywords: haemorroidal disease; haemorroidal crisis; internal haemorroids; external haemorroids; anal irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROCTOeze® PLUS (Experimental): Administration for 2 weeks of the MD PROCTOeze® PLUS to improve the haemorrhoidal symptomatology.
  Interventions: Device: Hydrophilic emulsion for the relief of haemorroidal symptoms

INTERVENTIONS:
Device: Hydrophilic emulsion for the relief of haemorroidal symptoms — Administration for 2 weeks of PROCTOeze® PLUS - a soft and light hydrophilic emulsion able to provide symptomatic relief of haemorrhoids and anal irritation.

SUMMARY:
This trial aims to evaluate the overall performance and safety of the MD PROCTOeze® PLUS in relieving symptomatology of haemorrhoidal disease and anal irritation in adult patients affected by Grade I-II (Goligher classification) haemorrhoids as assessed by the patient and the Investigator at the end of the treatment period.

DETAILED DESCRIPTION:
The protocol is based on what is already known on both the topic object of the study, i.e., the symptomatic treatment of haemorrhoids, and the investigational medical device - PROCTOeze® PLUS - which is a specific adjuvant for the symptomatic relief of internal and external haemorrhoids and anal irritation. Due to its formulation, it contributes to the physiological restoration of the anal and perianal tissues.

The tool used in this research is a PMCF, a procedure which, through a scientific method of detection (one or more questionnaires to be submitted to a representative sample of patients related to the issue of the research), allows to collect, and subsequently analyse, the data needed to study the relationships between different variables.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old.
* Patients diagnosed with Grade I - II symptomatic haemorrhoids (according to Goligher classification) confirmed by clinical and anoscopic or proctoscopic examination performed within 3 months before baseline.
* Patients able to do self-administration at home of the MD, for 14 days, to treat symptoms of haemorrhoids and anal irritation.
* Patient free from the following treatments for haemorrhoids for at least 4 weeks: laser treatments for haemorrhoids, steroidal or non-steroidal anti-inflammatory drugs, analgesics, any anti-haemorrhoidal treatment, anticoagulants, and antiplatelet agents.
* Patients able to communicate adequately with the Investigator and understand the tral questionnaire.
* Patients able to understand and who can provide valid informed consent to the trial.

Exclusion Criteria:

* Inflammatory and infectious disease of the digestive tract (e.g., IBD - Inflammatory Bowel Disease).
* Frequent hemorraidal bleeding
* Severe, uncontrolled hypertension, renal failure, cirrhosis, colorectal cancer, anal fissure or fistula.
* Patients with known sensitivity to the tested medical device or its components.
* Patients with any other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalisation during the study.
* Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Cristina Sisu, Dr., Principal Investigator — CMI Dr Sisu Lucia Cristina
Locations (1):
- C.M.I. Sisu Lucia Cristina, Craiova, Dolj, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start of enrolment (FPI) 5th November 2024; End of enrolment (LPI) 17th December 2024; End of treatment (LPO) 17th January 2025.
  Recruitment in the ambulatory of a General Physician office.
Groups:
- PROCTOeze® PLUS: Single arm, adults.
Period: Overall Study
Arm/Group | PROCTOeze® PLUS
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult patients affected by Grade I-II (Goligher classification) haemorrhoids that did not need hospitalization and treated as outpatients (the treatment will be self-administered at home).
Arm/Group | PROCTOeze® PLUS
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 50
Patients diagnosed with Grade I - II symptomatic haemorrhoids (Goligher classification) [Mean (Standard Deviation); unit: Score] — The Haemorrhoid Severity Score (HSS), a physician-reported outcome, will be completed by Investigator at baseline and day 30, at the end of the treatment with the medical device. Grades on a scale from 1 to 5, where lower grades are better with a total of 4 items on the questionnaire (minimum score 4, maximum score 20).
  The change of the total score of the HSS questionnaire between baseline and the end of the study will be assessed according to the Protocol by means of the Wilcoxon signed-rank test.
  Score | 8.50 (2.11)
Quality of Life measured by The Short Health Scale for Haemorrhoidal Disease (SHSHD) [Mean (Standard Deviation); unit: Score] — The Short Health Scale for Haemorrhoidal Disease (SHSHD) will be used to evaluate the Quality of Life. The questionnaire will be completed by the patient at baseline and day 30, at the end of the treatment with the medical device. Grades on a scale from 1 to 7, where lower grades are better, with a total of 4 items on the scale (minimum score 4, maximum score 28).
  The change of the total score of the SHSDH scale between baseline and the end of the study will be assessed according to the Protocol by means of the Wilcoxon signed-rank test.
  Score | 14.04 (7.79)
Quality of Life measured by The Haemorrhoidal Disease Symptom Score (HDSS) [Mean (Standard Deviation); unit: Score] — The Haemorrhoidal Disease Symptom Score (HDSS), a patient-reported outcome questionnaire, will be administered by Investigator to each patient at baseline and at day 30, at the end of the treatment with the medical device. Grades on a scale from 1 to 5, where lower grades are better, with a total of 5 items on the questionnaire (minimum score 5, maximum score 25).
  The change of the total score of the HDSS questionnaire between baseline and the end of the study will be assessed according to the Protocol by means of the Wilcoxon signed-rank test.
  Score | 10.12 (3.60)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Performance by the Improvement in the Quality of Life Measured Through the Score on The Short Health Scale for Haemorrhoidal Disease (SHSHD)
Description: The Short Health Scale for Haemorrhoidal Disease (SHSHD) will be used to evaluate the Quality of Life. The questionnaire will be completed by the patient at baseline and day 14, at the end of the treatment with the MD. Grades on a scale from 1 to 7, where lower grades are better, with a total of 4 items on the scale (minimum score 4, maximum score 28).
  Is an instrument with just 1 question in each of its 4 dimensions, including symptom burden, functional status, disease-specific worries, and general well-being measured according to A 7-point Likert scale to be summed giving a total score ranging from 4 to 28. The total of the four dimensions has been analyzed. The unit of measure is "score".
  SHS was adapted for HD (Short Health Scale for Haemorrhoidal Disease - SHSHD) in accordance with the Consensus-Based Standards for the Selection of Health Measurement Instruments (COSMIN) guidelines; SHSHD has shown to be a reliable and responsive measure for HRQoL.
Time Frame: From enrollment to the end of treatment on day 14.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | PROCTOeze® PLUS
Number analyzed (Participants) | 50
Score
  Baseline | 14.04 (7.79)
  End of Treatment | 7.80 (3.69)
Statistical Analysis 1: Comparison: PROCTOeze® PLUS; Test type: Superiority; p < 0.0001, Sign test; Mean difference (baseline - final) = 6.24, 28.2% CI 2-sided [4.67 to 7.81], Standard Deviation 5.51

2. Secondary Outcome: Assessment of Performance Through the Score on Haemorrhoid Severity Score (HSS) Reported by Physician
Description: HSS is a physician-reported measurement instrument based on PNR-Bleed classification. All four components in this classification system are graded into five grades ranging from 1 to 5. Grade 1 is the normal anal cushions and Grade 5 is the worst grade in a specific characteristic. HSS is the total score obtained by the sum of the numerical grades of all four characteristics of haemorrhoids in the PNR-Bleed classification. The minimum HSS score is 4 and the maximum score can be 20. The HSS score of a normal person without any signs and symptoms of haemorrhoids is 4. Calculation of the HSS helps in the quantification of the haemorrhoidal disease for further reference and is helpful in post-treatment patient follow-up to grade the response to treatment and to assess the effectiveness or failure of any particular treatment regimen for haemorrhoids.
  The total of the four dimensions has been analyzed. The unit of measure is "score".
Time Frame: From enrollment to the end of treatment on day 14.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | PROCTOeze® PLUS
Number analyzed (Participants) | 50
Score
  Baseline | 8.50 (2.11)
  End of treatment | 6.48 (2.17)
Statistical Analysis 1: Comparison: PROCTOeze® PLUS; Test type: Superiority; p < 0.0001, Sign test; Mean difference (baseline-final) = 2.02, 23.8% CI 2-sided [1.53 to 2.51], Standard Deviation 1.71

3. Secondary Outcome: Assessment of Performance Through the Score Haemorrhoidal Disease Symptom Score (HDSS) Reported by Patient
Description: The Haemorrhoidal Disease Symptom Score (HDSS), a patient-reported outcome questionnaire, will be administered by Investigator to each patient at baseline and at day 14, at the end of the treatment with the MD. Grades on a scale from 1 to 5, where lower grades are better, with a total of 5 items on the questionnaire.
  The HDSS is a patient-reported measurement instrument. It comprises five items. Symptoms are assessed using the patient-reported frequency of the 5 symptoms, including pain, itching, bleeding, soiling, and prolapse. Patients are instructed to answer based on their experience during the previous period. Each symptom is graded on a 5-point scale (0 = never, 1 = less than once a month, 2 = less than once a week, 3 = 1-6 days per week, 4 = every day or always), giving a total score ranging from 0 to 20.
  The total of the four dimensions has been analyzed. The unit of measure is "score".
Time Frame: From enrollment to the end of treatment on day 14.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | PROCTOeze® PLUS
Number analyzed (Participants) | 50
Score
  Baseline | 10.12 (3.60)
  End of treatment | 7.20 (2.47)
Statistical Analysis 1: Comparison: PROCTOeze® PLUS; Test type: Superiority; p < 0.0001, Sign test; Mean difference (baseline - final) = 2.92, 28.9% CI 2-sided [2.21 to 3.63], Standard Deviation 2.51

4. Secondary Outcome: Number of Treatment-emergent Adverse Events
Description: Safety and tolerability will be evaluated through the incidence of Adverse Event, Serious Adverse Event, Adverse Device Effect, Serious Adverse Device Effect, Anticipated Serious Adverse Device Effect, and Unanticipated Serious Adverse Device Effect assessed by Investigator and reported according to the current legislation for the whole study period. Device Deficiency will be also evaluated. The number of adverse events recorded will be evaluated to measure the safety of the MD.
Time Frame: From enrollment to the end of study on day 30.
Measure: Number; unit: Adverse events
Arm/Group | PROCTOeze® PLUS
Number analyzed (Participants) | 50
Adverse events | 0

ADVERSE EVENTS:
Time Frame: From enrollment up to end of follow-up, up to 30 days.
Arm/Group | PROCTOeze® PLUS
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
This study has no limitations since there are no drop-out patients and the symptoms measurements were performed with objective, widely-accepted and validated scales.

In addition, treatment compliance was optimal according to the patient diary, which was filled in daily during the treatment period by all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT06944951/Prot_SAP_ICF_000.pdf